CLINICAL TRIAL: NCT05471180
Title: Adjuvant Effect of Photobiomodulation in the Treatment of Incontinence-associated Dermatitis in Adults - a Randomized Controlled Clinical Trial
Brief Title: Adjuvant Effect of Photobiomodulation in the Treatment of Incontinence-associated Dermatitis in Adults
Acronym: DAI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The post graduated student change her project.
Sponsor: University of Nove de Julho (Other)
Collaborators: Adriana da Silva Magalhaes (Unknown)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, PhD, Postgraduate program professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dermatite
Record Dates: First submitted 2022-07-16; First posted 2022-07-22 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-07

CONDITIONS: Incontinence Associated Dermatitis; Diaper Rash; Photobiomodulation Therapy
Keywords: Incontinence associated dermatitis; Diaper Rash; Photobiomodulation therapy; Laser
MeSH Terms: conditions — Diaper Rash | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: participants who developed lesions that present erythema with intact skin and erythema with loss of continuity, resulting from IAD, will be included in the study. Participants will be randomly divided into 2 groups: Control group (n=39) - use of liquid protective film in spray + FBM simulation (placebo), Experimental group (n=39) - use of liquid protective film in spray + FBM. FBM will be performed with a 660 nm 100mW diode laser, 2 J per point, in 8 points and radiant exposure of 707 J/cm2. FBM will be applied once a day every 24 hours for 3 days in a row.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the researcher with a degree in Nursing, who will be responsible for carrying out the treatments (opening the envelopes of randomization), will know which treatment will be assigned to each participant (with photobiomodulation or its simulation). The researcher will not be involved in the assessment of injuries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Control group (n=39) - 3M Cavilon ® protective spray film + simulation of the use of laser (placebo) - after cleaning the skin, the pain scale will be applied and after application of FBM in the same points of the group that will undergo irradiation. To mimic the action of the laser, the BIP noise will be recorded and its activation will be done by the nursing employee who provides the care, after simulating the use of the laser, the use of the 3M Cavilon ® protective spray film will be applied. The application of the laser will be immediate in 8 points of the perineum region in the areas that present lesions, these applications will occur 1 x a day every 24 hours for three consecutive days. Skincare will be maintained with 3M Cavilon ® Cleansing Solution and the use of 3M Cavilon ® Protective Spray Film. A photographic record of the lesion will be made on days 0 and 3 of treatment and after 2 days after treatment to monitor the recovery of the IAD
  Interventions: Other: protective spray film
- Experimental group (Experimental): Experimental group (n= 39) 3M Cavilon ® protective spray film + FBM - skin cleaning and pain scale application will be performed and after laser application in 8 points of the affected perineum region, these applications will occur 1 x a day every 24 hours for three days. Skincare will be maintained with 3M Cavilon ® Cleansing Solution and the use of 3M Cavilon ® Protective Spray Film. The photographic record of the lesion will be performed on days 0 and 3, 5 and 7 days of treatment. To monitor the participants and observe the recovery and obtainment of skin healing. It will be used the Globaid tool that will be applied in both groups.
  Interventions: Other: protective spray film; Device: photobiomodulation therapy

INTERVENTIONS:
Other: protective spray film — Skincare will be maintained with 3M Cavilon ® Cleansing Solution and the use of 3M Cavilon ® Protective Spray Film.
Device: photobiomodulation therapy — application in 8 points of the affected perineum region, these applications will occur 1 x a day every 24 hours for three days.
  Arms: Experimental group

SUMMARY:
Incontinence-associated dermatitis (IAD) is an inflammation of the skin that occurs as a result of urine or feces contact on the perineal or perigenital region in adults. Lesions are typically located in the convex regions covered by diapers. The perineal region is the most affected, bringing pain and discomfort to the participant. The prevention and treatment of IAD must essentially follow two interventions: the control of incontinence/dampness and the implementation of a structured regimen of perineal care, seeking results for the restoration of skin integrity. Therefore, the gold standard for the treatment of IAD is skin hygiene, moisture control, and the use of a skin protector to restore skin integrity. Photobiomodulation has been used with excellent results in restoring skin integrity in acute and chronic wounds, but so far it has not been tested for IAD. To evaluate the effect of photobiomodulation in the treatment of incontinence-associated dermatitis in adults. A total of 78 with participant who developed lesions that present erythema with intact skin and erythema with loss of continuity, resulting from IAD, will be included in the study. Participants will be randomly divided into 2 groups: Control group use of liquid protective film in spray + FBM simulation (placebo), Experimental group (n=39) - use of liquid protective film in spray + FBM. FBM will be performed with a 660 nm 100mW diode laser, 2 J per point, in 8 points and radiant exposure of 707 J/cm2. FBM will be applied once a day every 24 hours for 3 days in a row. Both groups will continue with standard daily skin care and diaper changes every 3 hours. The primary endpoint was chosen for the 7-day IAD lesion cure rate study. A photographic record of the lesion area and measurements will be performed using a disposable ruler with the participant in a lithotomous position on the days of the evaluations. For the classification and characterization of the severity of IAD, the Ghent Global IAD Categorization tool will be applied. In addition, the size of the area will be analyzed using ImageJ software program. For pain assessment, the visual analog scale will be used in conscious participants and the BPS scale in participants with cognitive impairment and who are intubated. All outcomes will be evaluated at baseline, at 24 hours, 3 days, and 7 days.

DETAILED DESCRIPTION:
Incontinence-associated dermatitis (IAD) is an inflammation of the skin that occurs as a result of urine or feces contact on the perineal or perigenital region in adults. Lesions are typically located in the convex regions covered by diapers. The perineal region is the most affected, bringing pain and discomfort to the participant. The prevention and treatment of IAD must essentially follow two interventions: the control of incontinence/dampness and the implementation of a structured regimen of perineal care, seeking results for the restoration of skin integrity. Therefore, the gold standard for the treatment of IAD is skin hygiene, moisture control, and the use of a skin protector to restore skin integrity. Photobiomodulation has been used with excellent results in restoring skin integrity in acute and chronic wounds, but so far it has not been tested for IAD.

Materials and methods: A controlled, randomized, and blinded clinical study will be carried out on participants hospitalized in the Intensive Care sector, oncology, and coronary care unit of Hcor Associação Beneficente Síria. A total of 78 participants who developed lesions that present erythema with intact skin and erythema with loss of continuity, resulting from IAD, will be included in the study. Participants will be randomly divided into 2 groups: Control group (n=39) - use of liquid protective film in spray + FBM simulation (placebo), Experimental group (n=39) - use of liquid protective film in spray + FBM. FBM will be performed with a 660 nm 100mW diode laser, 2 J per point, in 8 points and radiant exposure of 707 J/cm2. FBM will be applied once a day every 24 hours for 3 days in a row. Both groups will continue with standard daily skin care and diaper changes every 3 hours. The primary endpoint was chosen for the 7-day IAD lesion cure rate study. A photographic record of the lesion area and measurements will be performed using a disposable ruler with the participant in a lithotomous position on the days of the evaluations. For the classification and characterization of the severity of IAD, the Ghent Global IAD Categorization tool will be applied. In addition, the size of the area will be analyzed using ImageJ software program. Pain will be assessed using a pain scale and a satisfaction questionnaire. All outcomes will be evaluated at baseline, at 24 hours, 3 days, and 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants or legal guardians who accept and fulfill the inclusion criteria for this study will sign the Free and Informed Consent Term (ICF) for authorization to participate in the study
* Adult subjects exposed to wet urine/stool or both, who have erythema in the perineal region with persistent erythema and skin loss according to the Ghent Global IAD Categorization Tool severity characterization scale in category 1 (1A) and category 2 (2A), without signs of infection
* Individuals of both male and female sex
* Individuals aged 21 or over

Exclusion Criteria:

* Individuals who do not have dermatitis in the perineal region, who have dermatitis
* Individuals classified by the Ghent Global IAD Categorisation Tool scale in Category 1-B who have persistent erythema with clinical signs of infection and Category 2-B) with skin loss with clinical signs of infection in the perineal region
* Instability such as arterial hypotension, respiratory discomfort that cannot be mobilized to perform the treatment of the lesion. Lesions in the perineal region with the presence of infection that requires the use of antibiotics, topical antifungals
* Individuals with serious injuries who benefit from treatments that will not be part of the conventional protocol
* Individuals who are pregnant
* Severity of injuries and signs of infections
* Individuals with skin lesions such as herpes in the perineal region
* Individuals with pressure injuries existing in the gluteal regions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
T- Healing rate of IAD lesion in 7 days | seventh day
  The participant will be evaluated by a calibrated member who will evaluate the participant with Globaid until the 7th day in which the lesion is expected to heal.

SECONDARY OUTCOMES:
Size of the lesion measured by its area | seventh day
  Size of the lesion measured by its area - A measurement of the lesion area will be made before the start of treatment on days 0 and 3 and day 7. To evaluate the lesion, the measurement in its greatest length and width will be considered, the measurements will be noted, and, later, multiplied one measurement by the other to obtain the area in cm²
Photographed for evaluation | seventh day
  The lesions will be photographed for evaluation on the 0th, 3rd, and 7th day and using the ImageJ® software "USA National Institutes of Health, Bethesda, MD ", analyses of the edge of each lesion will be performed, manually delimited with the mouse and the entire lesion will be circled for the calculation of the area, quantifying the total area of the lesions by the delimitation of the edges and, later, the dermatitis lesion index (ILD) will be calculated = (Initial area - Final area / Initial area), where ILD= 1 (100%) represents total revitalization; ILD=0 with no signs of revitalization; ILD>0 reductions and ILD. The computerized area of the lesion will be calculated by the scale in centimeters of the millimeter ruler photographed next to each lesion. This evaluation will be carried out by the same examiner who was not aware of the identification of the samples.
Ghent Global IAD Categorization Tool scale | seventh day
  The lesions will be photographed in a standardized way and will be evaluated by an experienced calibrated researcher, using the instrument for the evaluation of the Ghent Global IAD Categorization Tool scale from Globaid that characterizes the category of the lesion, individuals who do not have category 1 (1A) and category 2 (2A), demonstrate healing and wound healing. There are no signs of a cure if the category remains 1-(1A) and 2(2A). Individuals who evolve in category 1 (2B) and in category 2 (2B), will be considered as signs of severity, according to the scale and exit criteria of the study.
Pain assessment (Visual Analog Scale /Behavioral Pain Scale/ Pain Assessment in Advanced Dementia) | seventh day
  Pain assessment with the pain scale VAS with a score from 0 to 10 that will be applied to conscious participants who can inform the score of their pain,
  In intubated participants the Behavioral Pain Scale - BPS will be used with scores pain 0 to 12 in participants on mechanical ventilation, evaluating the following parameters: Facial expression, body movements, and Tolerance to mechanical ventilation the scale allows defining the pain intensity between 3 (no pain) and 12 (the greatest pain intensity).
  In adults with cognitive impairment, periods of confusion and dementia, the Pain Assessment in Advanced Dementia - PAINAD scale will be used, which has pain intensity from 0 to 10.The application of the scale will occur during intimate hygiene. Pain assessment will take place during intimate hygiene, which is the appropriate time to measure pain, this assessment will be done until the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina R Horliana, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We are planning to publish the protocol
Supporting Information: Study Protocol
Time Frame: 1 month
Access Criteria: everyone

REFERENCES:
- [Result] Bliss DZ, Funk T, Jacobson M, Savik K. Incidence and Characteristics of Incontinence-Associated Dermatitis in Community-Dwelling Persons With Fecal Incontinence. J Wound Ostomy Continence Nurs. 2015 Sep-Oct;42(5):525-30. doi: 10.1097/WON.0000000000000159. PMID 26336048
- [Result] Gray M, Black JM, Baharestani MM, Bliss DZ, Colwell JC, Goldberg M, Kennedy-Evans KL, Logan S, Ratliff CR. Moisture-associated skin damage: overview and pathophysiology. J Wound Ostomy Continence Nurs. 2011 May-Jun;38(3):233-41. doi: 10.1097/WON.0b013e318215f798. PMID 21490547
- [Result] Seifi B, Jalali S, Heidari M. Assessment Effect of Breast Milk on Diaper Dermatitis. Dermatol Reports. 2017 Mar 13;9(1):7044. doi: 10.4081/dr.2017.7044. eCollection 2017 Mar 13. PMID 28626535
- [Result] Gray M, Bliss DZ, Doughty DB, Ermer-Seltun J, Kennedy-Evans KL, Palmer MH. Incontinence-associated dermatitis: a consensus. J Wound Ostomy Continence Nurs. 2007 Jan-Feb;34(1):45-54; quiz 55-6. doi: 10.1097/00152192-200701000-00008. PMID 17228207
- [Result] Woo KY, Beeckman D, Chakravarthy D. Management of Moisture-Associated Skin Damage: A Scoping Review. Adv Skin Wound Care. 2017 Nov;30(11):494-501. doi: 10.1097/01.ASW.0000525627.54569.da. PMID 29049257
- [Result] Beeckman D, Van Damme N, Schoonhoven L, Van Lancker A, Kottner J, Beele H, Gray M, Woodward S, Fader M, Van den Bussche K, Van Hecke A, De Meyer D, Verhaeghe S. Interventions for preventing and treating incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2016 Nov 10;11(11):CD011627. doi: 10.1002/14651858.CD011627.pub2. PMID 27841440
- [Result] Beele H, Smet S, Van Damme N, Beeckman D. Incontinence-Associated Dermatitis: Pathogenesis, Contributing Factors, Prevention and Management Options. Drugs Aging. 2018 Jan;35(1):1-10. doi: 10.1007/s40266-017-0507-1. PMID 29243033
- [Result] Black JM, Gray M, Bliss DZ, Kennedy-Evans KL, Logan S, Baharestani MM, Colwell JC, Goldberg M, Ratliff CR. MASD part 2: incontinence-associated dermatitis and intertriginous dermatitis: a consensus. J Wound Ostomy Continence Nurs. 2011 Jul-Aug;38(4):359-70; quiz 371-2. doi: 10.1097/WON.0b013e31822272d9. PMID 21747256
- [Result] Kottner J, Blume-Peytavi U, Lohrmann C, Halfens R. Associations between individual characteristics and incontinence-associated dermatitis: a secondary data analysis of a multi-centre prevalence study. Int J Nurs Stud. 2014 Oct;51(10):1373-80. doi: 10.1016/j.ijnurstu.2014.02.012. Epub 2014 Feb 23. PMID 24636666
- [Result] Beeckman D, Van den Bussche K, Alves P, Arnold Long MC, Beele H, Ciprandi G, Coyer F, de Groot T, De Meyer D, Deschepper E, Dunk AM, Fourie A, Garcia-Molina P, Gray M, Iblasi A, Jelnes R, Johansen E, Karadag A, Leblanc K, Kis Dadara Z, Meaume S, Pokorna A, Romanelli M, Ruppert S, Schoonhoven L, Smet S, Smith C, Steininger A, Stockmayr M, Van Damme N, Voegeli D, Van Hecke A, Verhaeghe S, Woo K, Kottner J. Towards an international language for incontinence-associated dermatitis (IAD): design and evaluation of psychometric properties of the Ghent Global IAD Categorization Tool (GLOBIAD) in 30 countries. Br J Dermatol. 2018 Jun;178(6):1331-1340. doi: 10.1111/bjd.16327. Epub 2018 Apr 19. PMID 29315488
- [Result] Junkin J, Selekof JL. Beyond "diaper rash": Incontinence-associated dermatitis: does it have you seeing red? Nursing. 2008 Nov;38(11 Suppl):56hn1-10; quiz 56hn10-1. doi: 10.1097/01.NURSE.0000341725.55531.e2. PMID 19020456
- [Result] Chianca TC, Goncales PC, Salgado PO, Machado BO, Amorim GL, Alcoforado CL. Incontinence-associated dermatitis: a cohort study in critically ill patients. Rev Gaucha Enferm. 2017 Mar 30;37(spe):e68075. doi: 10.1590/1983-1447.2016.esp.68075. English, Portuguese. PMID 28380152
- [Result] Carr AN, DeWitt T, Cork MJ, Eichenfield LF, Folster-Holst R, Hohl D, Lane AT, Paller A, Pickering L, Taieb A, Cui TY, Xu ZG, Wang X, Brink S, Niu Y, Ogle J, Odio M, Gibb RD. Diaper dermatitis prevalence and severity: Global perspective on the impact of caregiver behavior. Pediatr Dermatol. 2020 Jan;37(1):130-136. doi: 10.1111/pde.14047. Epub 2019 Dec 2. PMID 31793090
- [Result] Burdall O, Willgress L, Goad N. Neonatal skin care: Developments in care to maintain neonatal barrier function and prevention of diaper dermatitis. Pediatr Dermatol. 2019 Jan;36(1):31-35. doi: 10.1111/pde.13714. Epub 2018 Dec 2. PMID 30506880
- [Result] Kajagar BM, Godhi AS, Pandit A, Khatri S. Efficacy of low level laser therapy on wound healing in patients with chronic diabetic foot ulcers-a randomised control trial. Indian J Surg. 2012 Oct;74(5):359-63. doi: 10.1007/s12262-011-0393-4. Epub 2012 Apr 11. PMID 24082586
- [Result] Maia ML, Bonjardim LR, Quintans Jde S, Ribeiro MA, Maia LG, Conti PC. Effect of low-level laser therapy on pain levels in patients with temporomandibular disorders: a systematic review. J Appl Oral Sci. 2012 Nov-Dec;20(6):594-602. doi: 10.1590/s1678-77572012000600002. PMID 23329239
- [Result] Gushiken LFS, Beserra FP, Bastos JK, Jackson CJ, Pellizzon CH. Cutaneous Wound Healing: An Update from Physiopathology to Current Therapies. Life (Basel). 2021 Jul 7;11(7):665. doi: 10.3390/life11070665. PMID 34357037
- [Result] Iryanov YM. Influence of Laser Irradiation Low Intensity on Reparative Osteogenesis and Angiogenesis Under Transosseous Osteosynthesis. J Lasers Med Sci. 2016 Summer;7(3):134-138. doi: 10.15171/jlms.2016.23. Epub 2016 Jul 18. PMID 28144431
- [Result] Hashmi JT, Huang YY, Osmani BZ, Sharma SK, Naeser MA, Hamblin MR. Role of low-level laser therapy in neurorehabilitation. PM R. 2010 Dec;2(12 Suppl 2):S292-305. doi: 10.1016/j.pmrj.2010.10.013. PMID 21172691
- [Result] Avci P, Gupta A, Sadasivam M, Vecchio D, Pam Z, Pam N, Hamblin MR. Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg. 2013 Mar;32(1):41-52. PMID 24049929